CLINICAL TRIAL: NCT01622244
Title: Coordinated Access to Care From Hospital Emergency Departments - Assessing Effectiveness and Cost-Effectiveness
Brief Title: Coordinated Access to Care From Hospital Emergency Departments
Acronym: CATCH-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: StMichael
Record Dates: First submitted 2012-06-04; First posted 2012-06-19 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2012-06

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Experimental): Participants will receive brief, intensive case management to connect them to health and social services and supports in the community
  Interventions: Other: Co-ordinated Access to Care from Hospital Emergency Departments; Other: Coordinated Access to Care from Hospital Emergency Departments
- Counseling and Resource Education (CARE) (Active Comparator): Participants will receive care as usual in the community. In addition, participants in this arm will receive an educational session and resource guide outlining available community-based services
  Interventions: Behavioral: Counseling and Resource Education

INTERVENTIONS:
Other: Co-ordinated Access to Care from Hospital Emergency Departments — brief, intensive case management for frequent users of hospital Emergency Departments who have mental health and/or addictions problems
  Arms: Intervention arm
Other: Coordinated Access to Care from Hospital Emergency Departments — Participants will receive brief, intensive case management to connect them to health and social services and supports in the community
  Arms: Intervention arm
Behavioral: Counseling and Resource Education — Participants will receive usual care as well as an educational session and resource guide outlining community-based services
  Arms: Counseling and Resource Education (CARE)

SUMMARY:
The study will assess the effectiveness and cost-effectiveness of providing brief, intensive case management for frequent users of hospital Emergency Departments who have mental health and/or addictions problems. The goals of the intervention are to support patients' transition to community-based health and social services and supports - including primary and urgent psychiatric care, peer support and other community services and supports - so as to improve patient wellbeing and reduce avoidable ED visits and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* legal adult status (age 18)
* able to give informed consent
* have made 5+ visits to participating hospital Emergency Department in the previous 12 months
* One of these visits will have been for a mental health and/or addiction problem.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Frequency of Emergency Department visits | Baseline, 6 and 12 months

SECONDARY OUTCOMES:
Changes in symptom severity | Baseline, 6 and 12 months
  A scales with good psychometric properties, the Colorado Symptom scale, will be used
Days in hospital | baseline, 6 and 12 months
Changes in substance use | baseline 6 and 12 months
  The Addiction Severity index will be used
Changes in health related quality of life | baseline, 6 and 12 months
  The SF-12 and EQ-5D will be used

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Stergiopoulos, MD, MHSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Stergiopoulos V, Gozdzik A, Tan de Bibiana J, Guimond T, Hwang SW, Wasylenki DA, Leszcz M. Brief case management versus usual care for frequent users of emergency departments: the Coordinated Access to Care from Hospital Emergency Departments (CATCH-ED) randomized controlled trial. BMC Health Serv Res. 2016 Aug 24;16(1):432. doi: 10.1186/s12913-016-1666-1. PMID 27557705